CLINICAL TRIAL: NCT02027948
Title: A Nutritional Management Algorithm in Older Patients With Locally Advanced Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-264
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Localized Stage I-III Esophageal Cancer; Gastroesophageal Junction Cancer
Keywords: nutritional management algorithm; nutritional and functional assessments; 13-264

ARMS (1):
- nutritional management (Experimental): The proposed study will be a prospective feasibility study of a nutritional management algorithm with risk-based guidelines in older adults (n=50) with newly diagnosed locally advanced esophageal cancer receiving preoperative or definitive chemoradiotherapy with an induction chemotherapy approach. Eligible patients must be age ≥ 65 years old. While all patients with esophageal cancer may benefit from this intervention, we wish to target the most vulnerable population (older patients who are at highest risk of malnutrition) in this pilot study.
  Interventions: Other: nutritional and functional assessments

INTERVENTIONS:
Other: nutritional and functional assessments — Patients will undergo nutritional & functional assessments along the continuum of their chemoradiotherapy treatment. The initial assessment will be measurements of height, weight, & baseline weight loss. Patients will receive chemotherapy & radiation as per standard practice at MSKCC, which is induction chemotherapy for approximately 3 weeks, followed by concurrent chemoradiotherapy. A commonly used regimen is weekly carboplatin (AUC 2) with paclitaxel (50 mg/m2) & radiation consisting of 5040 cGy over 28 fractions. Patients in this study will undergo assessments at three time points (at baseline, after induction chemotherapy, & post-treatment.) At baseline, all patients will complete the functional assessment, dysphagia scale, & Mini- Nutritional Assessment (MNA). According to the baseline MNA score, patients will be categorized as "normal nutrition," "at risk for malnutrition," or "malnourished" & receive the appropriate intervention.

SUMMARY:
Patients with esophageal and gastroesophageal junction (GEJ) cancer often have weight loss, swallowing problems, and poor appetite. This may affect their ability to tolerate cancer treatment.

The purpose of this study is to see if the researchers can apply a set of nutrition guidelines designed specifically for patients with cancer who are older than 65 years of age. The questions will allow them to assess the nutritional status and make appropriate referrals. If the patients are having swallowing problems or losing weight, the researchers want to address the nutritional problems early in the course of their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ age of 65; no maximum age limit.
* Patients who will receive induction chemotherapy followed by combined chemoradiotherapy at MSKCC for localized stage I-III esophageal or gastroesophageal junction cancer.
* Patients can receive chemoradiotherapy preoperatively prior to surgical resection or as definitive/primary chemoradiotherapy.
* Patients can be KPS ≥60, as long as primary provider feels that patient is candidate for combined modality chemoradiotherapy
* Be able to provide informed consent

Exclusion Criteria:

* Enrolled on a phase I trial
* Patients with a feeding tube previously placed.
* Not English-speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-12-23 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
feasibility of a nutritional management algorithm | 2 years
  Various validated assessments of nutritional status have been described. Nutritional status can be evaluated using: 1) anthropometric measures (i.e. weight loss, body mass index (BMI), triceps skin fold thickness, arm circumference), 2) immunological measurements (i.e. absolute lymphocyte count), and 3) serum protein markers (i.e. albumin, prealbumin, transferrin, and retinol-binding protein)

SECONDARY OUTCOMES:
treatment toxicity of chemoradiotherapy | 2 years
  Treatment toxicity of chemoradiotherapy will be summarized using descriptive statistics. Binomial proportions along with exact 95% confidence intervals will be estimated for proportions. Toxicity during the induction chemotherapy phase will be correlated with the baseline nutritional status (as determined by the MNA assessment) and baseline functional status using Fisher's exact test for categorical measures and Wilcoxon's rank sum test for numeric measures. Similarly, toxicity during chemoradiotherapy will be correlated with baseline MNA and functional status as well as with the malnutrition assessment using Fisher's exact test for categorical measures and Wilcoxon rank sum test for numeric measures.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Won, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk (Consent Only), Commack, New York
  - Memorial Sloan Kettering Cancer Center at Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering West Harrison (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/